CLINICAL TRIAL: NCT00659490
Title: A Randomised, Double Blind, Placebo-Controlled Study to Investigate the Analgesic Efficacy of a Single Dose of AZD1940, in Patients Undergoing Impacted Mandibular Third Molar Extraction
Brief Title: Study to Investigate the Analgesic Efficacy of a Single Dose of AZD1940
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3120C00006
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2010-05

CONDITIONS: Pain
Keywords: Analgesic effect; Molar extraction
MeSH Terms: conditions — Pain | interventions — N-(2-tert-butyl-1-((4,4-difluorocyclohexyl)methyl)-1H-benzo(d)imidazol-5-yl)ethanesulfonamide; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1940 (Experimental): AZD1940 800ug given predose
  Interventions: Drug: AZD1940
- Naproxen (Active Comparator): Naproxen 500mg given pre-surgery
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): Placebo given pre-surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1940 — 800ug oral administration
  Arms: AZD1940
Drug: Naproxen — 500mg oral administration
  Other Names: Naprosyn
  Arms: Naproxen
Drug: Placebo — Placebo given pre-surgery
  Arms: Placebo

SUMMARY:
The primary aim of this study is to investigate if AZD1940 can relieve the pain induced by the surgical removal of one lower wisdom-tooth. This will be done by comparing the effect of AZD1940 to placebo ("inactive substance") on pain. A number of patients will instead receive the common painkiller naproxen for comparison purposes. Rescue medication, acetaminophen, will be allowed if a need for additional painkillers would arise. A number of patients will receive Naproxen as control.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgical removal of one partial or complete impacted mandibular third molar.
* Provision of signed informed consent.
* Healthy males or non-fertile females.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives of the study, as judged by the investigator.
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorder, 4th edition.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, MD, Principal Investigator — Lifetree Clinical Research3838 South, 700 East, Suite 202Salt Lake City, Utah 84106, USA; Bror Jonzon, Study Chair — AstraZeneca R&D Södertälje, SE-151 85 Södertälje, Sweden
Locations (1):
- Research Site, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 centre (Lifetree Clinical Research, Salt Lake City, Utah, USA) recruited between Feb and May 2008
Pre-assignment Details: Screening for eligibility
Period: Overall Study
Arm/Group | AZD1940 | Placebo | Naproxen
Started | 61 | 59 | 31
Completed | 59 | 59 | 30
Not Completed | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1940 | Placebo | Naproxen | Total
Number analyzed (Participants) | 61 | 59 | 31 | 151
Age Continuous [Mean (Full Range); unit: Years] | 20.6 [18 to 35] | 21.0 [18 to 39] | 20.5 [18 to 35] | 20.7 [18 to 39]
Sex/Gender, Customized [Number; unit: Participants]
  Unknown | 61 | 59 | 31 | 151

OUTCOME MEASURES:

1. Primary Outcome: Pain Area Under the Curve 0-8h (AUC0-8h)
Description: Area under the Visual Analogue Scale (VAS, 0-100 mm) time curve 0-8h (from end of surgery). Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable.
Time Frame: 0-8 h(from end of surgery to 8 hours post surgery)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm*h
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm*h | 355 (182.3) | 356 (165.7) | 129 (105.4)

2. Secondary Outcome: Pain Area Under the VAS Versus Time Curve 0-4h (AUC0-4h)
Description: Area under the Visual Analogue Scale (VAS, 0-100 mm) time curve 0-4h (from end of surgery). Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable.
Time Frame: 0-4h (from end of surgery to 4 hours post surgery)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm*h
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm*h | 145 (93.5) | 143 (81.7) | 54 (45.0)

3. Secondary Outcome: Maximum Pain Based on VAS Scale
Description: Maximum pain recorded on a Visual Analogue Scale, VAS (0-100mm). Observed case.
  Maximum pain VAS (0-100mm, 0 = no pain - 100 = worst pain imaginable)
Time Frame: From end of surgery to 8h or time first intake of rescue medication (whichever came first)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm | 66 (24.5) | 65 (23.7) | 33 (20.7)

4. Secondary Outcome: Mean Pain Based on a VAS Scale
Description: Calculated as the area under the Visual Analogue Pain Scale (0-100 mm) versus time curve divided by time.Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable. Mean pain VAS (0-100mm, 0 = no pain - 100 = worst pain imaginable)
Time Frame: From end of surgery to 8h or time to first intake of rescue medication (whichever came first)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm | 31 (19.0) | 29 (16.7) | 13 (10.6)

5. Secondary Outcome: Pain at Jaw Movement AUC0-8h
Description: Area under the Visual Analogue Scale (VAS, 0-100 mm) of jaw movement versus time curve 0-8h (from end of surgery). Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable. Area under the curve 0-8h (from end of surgery) of VAS pain at jaw movement (0-100mm, 0 = no pain - 100 = worst pain imaginable)
Time Frame: 0-8h from end of surgery to 8 hours post surgery
Population: The analyses based on a per-protocol pop.
Measure: Mean (Standard Deviation); unit: mm*h
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm*h | 342 (192.0) | 337 (170.5) | 135 (119.7)

6. Secondary Outcome: Pain at Jaw Movement AUC0-4h
Description: Area under the Visual Analogue Scale (VAS, 0-100 mm) of jaw movement versus time curve 0-4h (from end of surgery). Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable. Area under the curve 0-4h (from end of surgery) of VAS pain at jaw movement (0-100mm0 = no pain - 100 = worst pain imaginable).
Time Frame: 0-4h after end of surgery to 4 hours post surgery
Population: The analyses based on a per-protocol pop.
Measure: Mean (Standard Deviation); unit: mm*h
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm*h | 142 (100.3) | 138 (86.9) | 53 (47.5)

7. Secondary Outcome: Maximum Pain at Jaw Movement
Description: Maximum pain at jaw movement recorded on a Visual Analogue Scale, VAS (0-100mm). Observed case.
  Maximum Pain at jaw movement VAS (0-100mm, 0 = no pain - 100 = worst pain imaginable)
Time Frame: From end of surgery to 8h or time to first intake of rescue medication (whichever came first)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm | 63 (25.2) | 63 (25.5) | 33 (24.7)

8. Secondary Outcome: Mean Pain at Jaw Movement
Description: Calculated as the area under the Visual Analogue Pain Scale (0-100 mm) of jaw movement versus time curve divided by time. Missing values in the pain-by-time curve was imputated using linear interpolation, last observation carried forward (LOCF) or first observation carried backwards (FOCB) as applicable. Mean Pain at jaw movement VAS (0-100mm, 0 = no pain - 100 = worst pain imaginable ).
Time Frame: From end of surgery to 8h or time to first intake of rescue medication (whichever came first)
Population: The analyses based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
mm | 32 (20.9) | 28 (16.9) | 14 (12.4)

9. Secondary Outcome: Pain at Rescue Medication
Description: Pain at time of first rescue medication (VAS 0-100mm). Only patients taking rescue are included in analysis. Observed case.
  Pain at time of first rescue medication (VAS 0-100mm, 0 = no pain - 100 = worst pain imaginable).
Time Frame: At time of first rescue medication taken before 8 hours after end of surgery
Population: Only patients taking rescue are included in analysis. The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 37 | 43 | 7
mm | 73 (20.6) | 70 (20.5) | 47 (13.8)

10. Secondary Outcome: Pain at Jaw Movement at Time of First Rescue Medication
Description: Pain at jaw movement at time of first rescue medication (VAS 0-100mm). Observed case.
  Pain at jaw movement at time of first rescue medication (VAS 0-100mm, 0 = no pain - 100 = worst pain imaginable).
Time Frame: At time of first rescue medication (before 8 hours after end on surgery)
Population: Only patients taking rescue are included in analysis. The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 37 | 43 | 7
mm | 67 (26.2) | 65 (25.5) | 53 (15.4)

11. Secondary Outcome: Time to First Intake of Rescue Medication.
Time Frame: From end of surgery to 8 hours following surgery
Population: Only patients actually taking rescue medication are included in analysis.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 37 | 43 | 7
Hours | 3.8 (1.05) | 3.7 (1.16) | 4.7 (1.18)

12. Secondary Outcome: Number of Patients Requesting Rescue Medication
Description: Observed case.
Time Frame: End of surgery up to 8hours following surgery
Population: The analyses are based on a per-protocol population.
Measure: Number; unit: Participants
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 61 | 59 | 31
Participants | 37 | 43 | 7

13. Secondary Outcome: Maximum Deterioration in Visual Analogue Mood Scale (VAMS) Stimulated
Description: Subjective qualities of mood in the subject are measured by letting the subject rate their subjective experiences of a number of adjectives using a series of visual analogue scales. Subjects are required to rate on 100-mm lines the extent to which they felt each adjective at a given time point from 'not at all' on the left end of the scale to 'extremely' on the right end of the scale. The VAMS commonly used in studies with cannabinoids consists of six adjectives and visual analogue scales: stimulated; high (as in drug high, elated); anxious; sedated; down (as in moody, depressed) and hungry.
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 41 | 12 | 28
mm | 22 (15.1) | 26 (23.9) | 28 (22.7)

14. Secondary Outcome: Maximum Deterioration in VAMS High
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 41 | 16 | 10
mm | 30 (25.2) | 12 (7.5) | 20 (22.8)

15. Secondary Outcome: Maximum Deterioration in VAMS Anxious
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 35 | 27 | 13
mm | 20 (20.0) | 15 (13.1) | 13 (15.1)

16. Secondary Outcome: Maximum Deterioration in VAMS Sedated
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 53 | 33 | 12
mm | 33 (24.8) | 21 (19.2) | 24 (26.4)

17. Secondary Outcome: Maximum Deterioration in VAMS Down
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included. The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 32 | 22 | 8
mm | 20 (20.4) | 25 (23.5) | 24 (29.0)

18. Secondary Outcome: Time to Max Deterioration in VAMS Stimulated
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 41 | 28 | 12
Minutes | 143 (94.9) | 163 (108) | 213 (190)

19. Secondary Outcome: Time to Max Deterioration in VAMS High
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 41 | 16 | 10
minutes | 115 (56.7) | 191 (180.0) | 193 (125.9)

20. Secondary Outcome: Time to Max Deterioration in VAMS Anxious
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 35 | 27 | 13
minutes | 126 (88.0) | 167 (115.7) | 212 (207.2)

21. Secondary Outcome: Time to Max Deterioration in VAMS Sedated
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 53 | 33 | 12
minutes | 190 (134.7) | 221 (134.5) | 227 (150.5)

22. Secondary Outcome: Time to Max Deterioration in VAMS Down
Description: as for outcome 13
Time Frame: Between dosing and 12h post-dose
Population: Only patients reporting a deterioration are included.The analyses are based on a per-protocol population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AZD1940 | Placebo | Naproxen
Number analyzed (Participants) | 32 | 22 | 8
minutes | 227 (156.2) | 262 (106.3) | 349 (243.3)

ADVERSE EVENTS:
Arm/Group | AZD1940 | Placebo | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59 | 0/31
Other Adverse Events (participants affected / at risk) | 3/61 | 2/59 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1940 (N=61) | Placebo (N=59) | Naproxen (N=31)
Presyncope, Syncope (Nervous system disorders) | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has exclusive rights to publish the results of the tudy